CLINICAL TRIAL: NCT00181597
Title: A Phase II Study of Trilostane for Androgen-Independent Prostate Cancer
Brief Title: Trilostane for Androgen-Independent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-037
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: Trilostane; Androgen-independent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — trilostane; Hydrocortisone

INTERVENTIONS:
Drug: Trilostane — Taken orally once a day for three days then twice daily thereafter.
Drug: Hydrocortisone — Taken orally with trilostane.

SUMMARY:
The main purpose of this study is to test the safety of trilostane by looking at what effects, good and bad, it has on patients with androgen-independent prostate cancer.

DETAILED DESCRIPTION:
* Patients will take trilostane orally once a day for three days, then twice a day thereafter.
* Patients will complete a daily drug log recording the date, time and number of capsules taken.
* Trilostane may moderately decrease the production of steroids by the adrenal glands. In order to prevent any symptoms related to decreased steroid production, patients will also take hydrocortisone at the same time as the trilostane.
* While the patients are on treatment blood work will be done after 2 weeks and then every 4 weeks to test the levels of PSA in the blood. On weeks 4 and 8 of treatment additional blood work will be done to check hormone levels. Blood pressure and pulse rate will also be taken every 4 weeks.
* Depending upon disease status, radiological testing (CT scan, x-rays, and/or bone scan) may be repeated every 12 weeks.
* Patients will remain on study treatment as long as their disease responds and they do not experience any severe side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma
* Disease progression despite androgen depravation therapy and antiandrogen withdrawal
* Progressive measurable disease or bone scan progression or PSA progression
* Serum total testosterone < 50ng/ml
* Creatinine < 2.0 mg/dl
* ALT < 2 x ULN
* CALGB performance status of 0,1, or 2

Exclusion Criteria:

* Radiation therapy within 4 weeks
* Antiandrogen within 8 weeks
* Other secondary hormonal therapy or investigational agents within 4 weeks
* Prior chemotherapy for androgen-independent prostate cancer
* History of adrenal insufficiency
* Known brain metastases
* Severe liver or renal disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-03; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
activity of trilostane in men with androgen-independent prostate cancer. | 4 years

SECONDARY OUTCOMES:
serum levels of gonadal and adrenal steroids | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts